CLINICAL TRIAL: NCT06987058
Title: An Open-label Multicenter Rollover Study to Provide Continued Treatment to Participants Previously Enrolled in a RVU120 Clinical Study
Brief Title: RVU120 Rollover Study
Acronym: ROVER-01
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ryvu Therapeutics SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROVER-01; 2025-521673-14-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors; Acute Myeloid Leukaemia (AML); High-risk Myelodysplastic Syndrome
Keywords: Relapse; Refractory; Metastatic; Advanced; Solid Tumor; AML; Myelodysplastic syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence; Neoplasm Metastasis; Myelodysplastic Syndromes

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RVU120 single agent (Experimental): Study intervention is assigned in accordance with the parent protocol and consists of RVU120-based treatment.
  Interventions: Drug: RVU120

INTERVENTIONS:
Drug: RVU120 — RVU120 is a potent, selective inhibitor of CDK8 and its paralog CDK19
  Other Names: SEL120

SUMMARY:
This is a multicenter rollover study to provide continued treatment to eligible participants previously enrolled in a RVU120 clinical study and to evaluate the safety of the treatment and record the time on treatment when continued under the same regimen as in the parent study.

To be eligible for this rollover study, participants must be continuing to benefit from their treatment, show an acceptable safety profile, and not have access to commercially available comparator anticancer therapy. Once transitioned to this study, participants will continue with their next planned dose per the regimen of their parent study.

DETAILED DESCRIPTION:
Participants may continue treatment until loss of clinical benefit as judged by the investigator, unacceptable toxicity, start of subsequent anticancer therapy, or until any other criterion for withdrawal from the treatment or the study is met.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is enrolled in a RVU120 clinical study and receiving RVU120-based treatment given alone or in combination for at least 5 cycles.
2. The participant is currently benefiting from, and expected to continue to benefit from, RVU120-based treatment according to the criteria set out in the parent study protocol and according to the judgment of the investigator and sponsor.
3. The participant does not have access to commercially available comparator anticancer therapy.
4. Contraceptive use by participants or participant partners should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
5. The participant signed the rollover study ICF prior to any study-related procedure or study data collection.
6. The participant agrees not to donate blood during study participation and until 28 weeks (~6.5 months) after the last dose.
7. The investigator considers the participant to be eligible for participation in the rollover study.

Exclusion Criteria:

1. Presence of toxicity that cannot be adequately managed.
2. Concurrent participation in any therapeutic clinical study other than the parent study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (Safety and Tolerability) | 12 months
  Number and grade of adverse events assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Duration of response | 12 months
  Time from the first administration of RVU120-based treatment in the parent study until discontinuation of RVU120-based treatment for any reason in the rollover study.

CONTACTS AND LOCATIONS:
Locations (2):
- Uniwersyteckie Centrum Kliniczne, Gdansk, Poland
- Clinica Universidad de Navarra, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: No